CLINICAL TRIAL: NCT06545240
Title: Performance of Mid-Upper Arm Circumference for Detection of Severe Acute Malnutrition in Indonesian Under-Fives
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Klara Yuliarti, Principal Investigator, Indonesia University
Other Study IDs: 19-12-1452
Record Dates: First submitted 2024-07-31; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Severe Acute Malnutrition
Keywords: mid-upper arm circumference; sensitivity; severe acute malnutrition; specificity; WHZ index
MeSH Terms: conditions — Severe Acute Malnutrition; Hypersensitivity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mid-upper arm circumference — Mid-upper arm circumference was taken using non-stretchable band SECA 202
  Other Names: Weight measurement; Length and height measurement

SUMMARY:
WHO recommends 11.5 cm as a cut-off point of Mid-Upper Arm Circumference (MUAC) to detect and/or diagnose severe acute malnutrition (SAM) in under-five. MUAC is practical and useful, especially in area with limited facilities which has no standardized scale and infantometer. However, several studies showed that this cut-off need to be evaluated as it has modest detection rate for SAM. This study aims to evaluate diagnostic value of MUAC with 11.5 cm cut-off compared to WHZ as gold standard to identify SAM. The sensitivity, specificity, positive and negative predictive value of MUAC with 11.5 cm as a standard cut-off will be evaluated.

This study also aim to find new cut-off value that may offer better diagnostic performance. The main research questions were:

What is the diagnostic accuracy of Mid-Upper Arm Circumference (MUAC) compared to the Weight for Height Z Score (WHZ) in identifying SAM in children, and what is the optimal MUAC cut-off value for enhanced diagnostic performance?

ELIGIBILITY:
Inclusion Criteria:

* under-fives that 6-59 months-old

Exclusion Criteria:

* ascites
* edema
* hydrocephalus
* tumor or oncologic diseases
* organomegaly
* uncooperative during measurement

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study was conducted in the largest primary community health care facility in Cengkareng Jakarta and have 29.110 registered under-fives in its service area.
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Diagnostic value of MUAC in diagnosing SAM compare to WHZ-index | 2 months
  To evaluate sensitivity, specificity, positive and negative predictive value of MUAC

SECONDARY OUTCOMES:
Finding new cut off value that offer better diagnostic performance using ROC | 2 months
  To compare sensitivity, specificity, positive and negative predictive value of MUAC with 11.5 cm as standard cut off and to new cut-off value that may offer better diagnostic performance

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Puskesmas Cengkareng, Jakarta, DKI Jakarta
  - RSUPN Dr Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta

IPD SHARING:
Plan to Share IPD: No